CLINICAL TRIAL: NCT03263819
Title: POSTURAL ORTHOSTATIC TACHYCARDIA SYNDROME AND GASTROINTESTINAL SYMPTOMS: Contribution of Gastrointestinal Peptides
Brief Title: Gastrointestinal Symptoms in Postural Orthostatic Tachycardia Syndrome
Acronym: POTS-GUT
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 170052
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Postural Tachycardia Syndrome
Keywords: gastrointestinal hormones; Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be retain for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POTS: Postural Tachycardia Syndrome: patients with postural orthostatic tachycardia syndrome diagnosis.
  Interventions: Diagnostic Test: Oral glucose tolerance test
- Healthy controls: Patients with Postural orthostatic tachycardia syndrome who has peripheral neuropathy
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — 75 grams of glucose

SUMMARY:
Patients with POTS experience significant gastrointestinal symptoms. Current evidence suggesting that abnormal post-ganglionic sympathetic function could play a role in the pathophysiology of these GI abnormalities. Sympathetic fiber regulate motor and the postprandial GI peptides secretion.

The focus of the present proposal is to determine glucose homeostasis, GI motility, and their association with GI and cardiovascular symptoms in POTS patients versus healthy controls. Furthermore, we will determine differences in these outcomes in POTS patients with and without evidence of postganglionic sympathetic fiber neuropathy.

As a long-term goal, this study can lead us to understand the pathophysiology of common co-morbidities in patients with POTS to provide new treatment approaches and prevention strategies.

DETAILED DESCRIPTION:
Postural Tachycardia Syndrome (POTS) is a disabling condition that mostly affects young women in their reproductive age. It is characterized by chronic (>6 months) orthostatic intolerance symptoms (palpitation, lightheadedness, blurred vision and mental clouding) triggered by assuming an upright posture and that improved upon recumbency. These symptoms are associated with a rapid increase in heart rate (≥30 bpm) that occur within 10 minutes upon standing. POTS is estimated to affect up to 3 million persons in the United States and is considered a syndrome rather than a single disease.

The pathophysiology of POTS is complex, and are related to abnormal cardiovascular autonomic adaptation to postural changes. Under normal conditions, the assumption of upright posture does not result in major changes in blood pressure due to the integration of complex autonomic, circulatory and neurohumoral responses. Upright posture-induced a fluid shift of approximately 700 mL of blood from the upper thorax to the splanchnic circulation and lower extremities, which result in decrease in venous return to the heart, ventricular filling, and stroke volume. These changes cause unloading of the arterial baroreceptors and increase in sympathetic activity, vasoconstriction and restoration of stroke volume and cardiac output.

In POTS patients, multiple mechanisms have been proposed to explain the exaggerated increase in heart rate. The orthostatic tachycardia could be a compensatory phenomenon to hypovolemia, impaired sympathetic-mediated vasoconstriction or increased vascular compliance. The later could induce an exaggerated fluid shift upon standing from thorax to lower body. Depending on the mechanism involved different POTS phenotype has been described: (i) hypovolemic POTS; (ii) neuropathic POTS; and (iii) POTS associated with Ehlers-Danlos and joint hypermobility syndrome (EDS/JHS). Of note, there is overlapping in the pathophysiology of POTS with patients having more than one etiology.

In addition to the cardiovascular symptoms, patients with POTS experience significant gastrointestinal symptoms namely nausea, bloating, diarrhea or even severe constipation. Furthermore, large meals or high carbohydrate meals exacerbates the feelings of palpitations, weakness, and fatigue in these patients.

Multiple studies have reported the presence of alterations in the gastrointestinal motility. Pooled data from 352 patients recruited from 6 different studies, showed 21-80% prevalence of nausea, vomiting, and abdominal pain. In four of these studies that measured gastric motility, they found that 43% prevalence of rapid gastric emptying and 20% prevalence of delayed gastric emptying. Furthermore, Al-Shekhlee et al. reported a high prevalence of impaired sudomotor function in the POTS patients who reported GI symptoms suggesting that abnormal post-ganglionic sympathetic function could play a role in the pathophysiology of these GI abnormalities.

We previously defined a subgroup of POTS patients in whom we detected a partial peripheral autonomic neuropathy primarily affecting lower extremities (neuropathic POTS). These subjects had decreased norepinephrine spillover in response to sympathetic activation and abnormal sweat volumes and prolonged latency detected by quantitative sudomotor axon reflex (QSART). Recently, Gibbons and Freeman (2013) strengthen the definition by providing histological evidence of neuronal damage with the inclusion of skin biopsies with specific staining for autonomic dense fiber and sensitivity assessment.

In Neuropathic POTS there is evidence of impaired vasomotor tone in different specific vascular bed, particularly the splanchnic circulation. Tani et al. reported reduced splanchnic vascular resistance and increase in resting mesenteric blood flow providing evidence of splanchnic denervation.

In summary, there is evidence of post-ganglionic sympathetic denervation is a subset of patients with POTS. The most current definition are based on the presence of abnormal sudomotor and sensitivity assessment.

The sympathetic nervous system (SNS) provide innervation to the enteric ganglia, the circular muscles of sphincters, and the mucosa of the stomach and intestines. The SNS also negatively regulate the motor and secretory functions of the gastrointestinal (GI) tract. Browning and Travagli (2014) reported that the absence of sympathetic inhibitory innervation causes excessive and uncoordinated activity in the GI tract. Indicating that a preserved ANS (autonomic nervous system) regulation of the GI tract is crucial for the maintenance of normal GI motility.

In addition to regulating the motor function, the SNS and parasympathetic nervous system (PNS) regulate the postprandial GI peptides secretion by enteroendocrine cells (EEC). EECs are the first line components of the Brain-Gut axis. Multiple peptides, such as incretins (GLP-1, GLP-2, GIP), and PYY (peptide YY) are important for the maintenance of glucose homeostasis. They are secreted by a different type of EEC in the GI tract. Prior to their absorption, nutrients in the GI lumen are important stimuli for peptide secretion in the ileum in rats, pigs , and humans. These peptides are secreted before the bulk of ingested meal reaches to the ileum, suggesting the presence of a neuronal/endocrine pathway in GI tract.

In summary, the SNS through innervation the gut smooth muscle; ENS (enteric nervous system) and EECs negatively regulate the GI motor function and incretins secretion which impact glucose homeostasis.

Evidence from animal models showed that when rats underwent removal of the superior autonomic mesenteric ganglia that contains mostly SNS neurons and were challenged with an oral glucose gavage; plasma insulin and C-peptide secretion were increased compared with controls (non-ganglionectomised rats). Furthermore, glucose levels were much lower in the ganglionectomised rats suggesting that the SNS splanchnic innervation plays a critical role in the maintenance of glucose homeostasis. The increased secretion of insulin and C-peptide levels in this model could be explained by an increase in incretin hormonal release. Additional studies using isolated guineas pig ileum (in vitro model) showed that GLP-1 secretion is inhibited by SNS nerve stimulation which is mediated by α-adrenergic receptors.

In summary, in the absence of sympathetic tone on ENS and EECs the incretins secretion increases which may cause low levels of plasma glucose.

The focus of the present proposal is to determine glucose homeostasis, GI motility, and their association with GI and cardiovascular symptoms in POTS patients versus healthy controls. Furthermore, we will determine differences in these outcomes in POTS patients with and without evidence of postganglionic sympathetic fiber neuropathy.

The glucose homeostasis will be evaluated by a modified oral glucose tolerance test (OGTT). In addition, we will assess GI symptoms and hemodynamics before and after oral glucose (at minute 0, 30, 60, 90, and 120). The plasma levels of GI peptides (GLP-1, GLP-2, PYY, glucagon, C-peptide, insulin) will be measured in different time points after oral glucose. Gastric emptying will be evaluated by acetaminophen absorption test (AAT). The LPS (lipopolysaccharide), LBP (lipopolysaccharid-binding protein), sCD14, and I-FABP (faty acid-binding protein) as GUT cells damage markers will be measured at baseline. The following technics will be used in this study:

1. Oral glucose tolerance test (OGTT): In the case of OGTT, subjects will be given a ready-to-use test solution (TRUTOL® 75, Thermo Scientific, USA) containing 75 g glucose dissolved in 300 mL water, immediately after fasting blood sampling. They will be instructed to drink the test solution within 5 mins. Blood samples will be drawn at 5, 10, 15, 30, 60, 90, and 120 minutes after drinking the ready-to-use test solution. Gastric emptying will be measured by acetaminophen absorption test.
2. Acetaminophen absorption test (AAT): Acetaminophen (20 mg/kg) will be given to patients. Serum acetaminophen will be determined by fluorescence polarization immunoassay. This assay uses a six-point calibration curve, and the detection limit is 4 µmol/L. The coefficient of variation is less than 5%. Estimation of the rate of gastric emptying was based on serum concentrations of acetaminophen in the blood samples collected. An algorithm that transforms serum concentrations of paracetamol into estimates of gastric emptying was applied. This algorithm adjusts for first-pass metabolism, unequal distribution and individual rate of elimination, and provides estimates for the percentage of meal emptied from the stomach as a function of time.
3. Gastrointestinal symptoms scoring: The 2-page questionnaire is based on elements from a questionnaire that have been validated with some modifications. The questionnaire contains 17 questions on the frequency of GI symptoms that have been troublesome in the preceding 6 months. The frequency of each symptom is rated on seven-point Likert scale from no discomfort to very severe discomfort.
4. Hemodynamic symptoms scoring: Hemodynamic symptoms will be measured by using the Vanderbilt POTS Symptom Score. The patients will be asked to rate the severity of 9 symptoms on a 0-10 scale (with 0 reflecting an absence of symptoms). The sum of the scores at each time point will be used as a measure of symptom burden. The 9 symptoms are: mental clouding, blurred vision, shortness of breath, rapid heartbeat, tremulousness, chest discomfort, headache, lightheadedness, and nausea. This symptom score has been previously used by our center, and the symptoms were chosen as they reflect common complaints of patients with POTS.
5. Glucose and insulin levels: Glucose levels will be measured with a glucose analyzer (YSI Life Sciences, Yellow Springs, OH).
6. GI peptides measurements: The plasma designated for GLP-1 measurement will be supplemented with aprotinin (1,000 kallikrein inactivation unit (KIU)/ml) and dipeptidyl peptidase-4 inhibitor (20 μl/ml plasma; Millipore, St. Charles, MO). Plasma insulin, c-peptide, glucagon, GIP, active GLP-1 (7-37 and 7-36 amide), peptide YY, pancreatic polypeptide, and leptin were measured by multiplex immunoassays (Luminex, Millipore).

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Postural Tachycardia Syndrome: Heart rate increase >30 bpm from supine within 10 min of standing, in the absence of orthostatic hypotension (>20/10 mmHg fall in blood pressure), with chronic symptoms (> 6 months), and in the absence of other acute cause of orthostatic tachycardia.
* Able and willing to provide informed consent
* Female premenopausal subjects must utilize adequate birth control and willingness to undergo serum beta-hCG (human chorionic gonadotropin) testing

Exclusion Criteria:

* Use of acetaminophen or acetaminophen-related drugs (over-the-counter) in the 24 hours prior to the study.
* Hypertension (>150 mmHg systolic and >100 mmHg diastolic) based on history or findings on screening.
* Orthostatic hypotension (consistent decrease in BP >20/10 mmHg with 10 min stand)
* Pregnancy
* History of type 1 or type 2 diabetes mellitus
* Cardiovascular disease, such as myocardial infarction within 6 months, angina pectoris, significant arrhythmia (sinus tachycardia is not excluded), deep vein thrombosis, pulmonary embolism
* History of serious neurologic disease
* Impaired hepatic function (aspartate amino transaminase and/or alanine amino transaminase >1.5 x upper limit of normal range)
* Impaired renal function (serum creatinine >1.5 mg/dL)
* Hematocrit <28%
* Any underlying or acute disease requiring regular medication that could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Inability to comply with the protocol

Healthy control subjects

Defined as subjects without any significant past medical history, non-smokers, and on no chronic medications at the time of the study. Healthy control subjects will be age- and BMI-matched to the POTS patients.

Positive control

Patients with complete autonomic neuropathy (pure autonomic failure) will be enrolled as positive control. This condition is defined as complete autonomic failure based on AFT (autonomic function test) and norepinephrine plasma levels less than 100 pg/ml.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: The participants with POTS and "complete autonomic failure" will be recruited from patients referred to the Vanderbilt University Autonomic Dysfunction Center. Additional patients will be recruited from the POTS registry in ResearchMatch, and information about the study will be posted on websites associated with POTS support groups. Healthy volunteers will be recruited from a population of previous participants in autonomic studies, through the ResearchMatch.org database, Subject Locator, and through advertising and emails around the Vanderbilt community.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: cyndya shibao, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal AK, Garg R, Ritch A, Sarkar P. Postural orthostatic tachycardia syndrome. Postgrad Med J. 2007 Jul;83(981):478-80. doi: 10.1136/pgmj.2006.055046. PMID 17621618
- [Background] Postural Tachycardia Syndrome Information Page: National Institute of Neurological Disorders and Stroke (NINDS) [Internet]. [cited 2016 Aug 15]. Available from: http://www.ninds.nih.gov/disorders/postural_tachycardia_syndrome/postural_tachycardia_syndrome.htm
- [Background] Dysautonomia International: Postural Orthostatic Tachycardia Syndrome [Internet]. [cited 2016 Aug 15]. Available from: http://www.dysautonomiainternational.org/page.php?ID=30
- [Background] Zhang Q, Chen X, Li J, Du J. Clinical features of hyperadrenergic postural tachycardia syndrome in children. Pediatr Int. 2014 Dec;56(6):813-816. doi: 10.1111/ped.12392. Epub 2014 Oct 15. PMID 24862636
- [Background] Mathias CJ, Low DA, Iodice V, Owens AP, Kirbis M, Grahame R. Postural tachycardia syndrome--current experience and concepts. Nat Rev Neurol. 2011 Dec 6;8(1):22-34. doi: 10.1038/nrneurol.2011.187. PMID 22143364
- [Background] Lawal A, Barboi A, Krasnow A, Hellman R, Jaradeh S, Massey BT. Rapid gastric emptying is more common than gastroparesis in patients with autonomic dysfunction. Am J Gastroenterol. 2007 Mar;102(3):618-23. doi: 10.1111/j.1572-0241.2006.00946.x. PMID 17100966
- [Background] Antiel RM, Risma JM, Grothe RM, Brands CK, Fischer PR. Orthostatic intolerance and gastrointestinal motility in adolescents with nausea and abdominal pain. J Pediatr Gastroenterol Nutr. 2008 Mar;46(3):285-8. doi: 10.1097/MPG.0b013e318145a70c. PMID 18376245
- [Background] Wang LB, Culbertson CJ, Deb A, Morgenshtern K, Huang H, Hohler AD. Gastrointestinal dysfunction in postural tachycardia syndrome. J Neurol Sci. 2015 Dec 15;359(1-2):193-6. doi: 10.1016/j.jns.2015.10.052. Epub 2015 Oct 30. PMID 26671111
- [Background] Loavenbruck A, Iturrino J, Singer W, Sletten DM, Low PA, Zinsmeister AR, Bharucha AE. Disturbances of gastrointestinal transit and autonomic functions in postural orthostatic tachycardia syndrome. Neurogastroenterol Motil. 2015 Jan;27(1):92-8. doi: 10.1111/nmo.12480. Epub 2014 Dec 6. PMID 25483980
- [Background] Park KJ, Singer W, Sletten DM, Low PA, Bharucha AE. Gastric emptying in postural tachycardia syndrome: a preliminary report. Clin Auton Res. 2013 Aug;23(4):163-7. doi: 10.1007/s10286-013-0193-y. Epub 2013 May 25. PMID 23708963
- [Background] Al-Shekhlee A, Lindenberg JR, Hachwi RN, Chelimsky TC. The value of autonomic testing in postural tachycardia syndrome. Clin Auton Res. 2005 Jun;15(3):219-22. doi: 10.1007/s10286-005-0282-7. PMID 15944872
- [Background] Lomax AE, Sharkey KA, Furness JB. The participation of the sympathetic innervation of the gastrointestinal tract in disease states. Neurogastroenterol Motil. 2010 Jan;22(1):7-18. doi: 10.1111/j.1365-2982.2009.01381.x. Epub 2009 Aug 14. PMID 19686308
- [Background] Browning KN, Travagli RA. Central nervous system control of gastrointestinal motility and secretion and modulation of gastrointestinal functions. Compr Physiol. 2014 Oct;4(4):1339-68. doi: 10.1002/cphy.c130055. PMID 25428846
- [Background] Mundinger TO, Cummings DE, Taborsky GJ Jr. Direct stimulation of ghrelin secretion by sympathetic nerves. Endocrinology. 2006 Jun;147(6):2893-901. doi: 10.1210/en.2005-1182. Epub 2006 Mar 9. PMID 16527847
- [Background] Moran GW, Leslie FC, Levison SE, Worthington J, McLaughlin JT. Enteroendocrine cells: neglected players in gastrointestinal disorders? Therap Adv Gastroenterol. 2008 Jul;1(1):51-60. doi: 10.1177/1756283X08093943. PMID 21180514
- [Background] Roberge JN, Brubaker PL. Regulation of intestinal proglucagon-derived peptide secretion by glucose-dependent insulinotropic peptide in a novel enteroendocrine loop. Endocrinology. 1993 Jul;133(1):233-40. doi: 10.1210/endo.133.1.8319572.
- [Background] Knapper JM, Heath A, Fletcher JM, Morgan LM, Marks V. GIP and GLP-1(7-36)amide secretion in response to intraduodenal infusions of nutrients in pigs. Comp Biochem Physiol C Pharmacol Toxicol Endocrinol. 1995 Jul;111(3):445-50. doi: 10.1016/0742-8413(95)00046-1. PMID 8564784
- [Background] Layer P, Holst JJ, Grandt D, Goebell H. Ileal release of glucagon-like peptide-1 (GLP-1). Association with inhibition of gastric acid secretion in humans. Dig Dis Sci. 1995 May;40(5):1074-82. doi: 10.1007/BF02064202. PMID 7729267
- [Background] Blat S, Guerin S, Chauvin A, Seve B, Morgan L, Cuber JC, Malbert CH. The vagus is inhibitory of the late postprandial insulin secretion in conscious pigs. Auton Neurosci. 2002 Oct 31;101(1-2):68-77. doi: 10.1016/s1566-0702(02)00184-4. PMID 12462361
- [Background] Orskov C, Rabenhoj L, Wettergren A, Kofod H, Holst JJ. Tissue and plasma concentrations of amidated and glycine-extended glucagon-like peptide I in humans. Diabetes. 1994 Apr;43(4):535-9. doi: 10.2337/diab.43.4.535. PMID 8138058
- [Background] Kumakura A, Shikuma J, Ogihara N, Eiki J, Kanazawa M, Notoya Y, Kikuchi M, Odawara M. Effects of celiac superior mesenteric ganglionectomy on glucose homeostasis and hormonal changes during oral glucose tolerance testing in rats. Endocr J. 2013;60(4):525-31. Epub 2013 Jan 11. PMID 23318598
- [Background] Hansen L, Lampert S, Mineo H, Holst JJ. Neural regulation of glucagon-like peptide-1 secretion in pigs. Am J Physiol Endocrinol Metab. 2004 Nov;287(5):E939-47. doi: 10.1152/ajpendo.00197.2004. PMID 15475512
- [Background] Jacob G, Costa F, Shannon JR, Robertson RM, Wathen M, Stein M, Biaggioni I, Ertl A, Black B, Robertson D. The neuropathic postural tachycardia syndrome. N Engl J Med. 2000 Oct 5;343(14):1008-14. doi: 10.1056/NEJM200010053431404. PMID 11018167
- [Background] Schondorf R, Low PA. Idiopathic postural orthostatic tachycardia syndrome: an attenuated form of acute pandysautonomia? Neurology. 1993 Jan;43(1):132-7. doi: 10.1212/wnl.43.1_part_1.132. PMID 8423877
- [Background] Gibbons CH, Bonyhay I, Benson A, Wang N, Freeman R. Structural and functional small fiber abnormalities in the neuropathic postural tachycardia syndrome. PLoS One. 2013 Dec 27;8(12):e84716. doi: 10.1371/journal.pone.0084716. eCollection 2013. PMID 24386408
- [Background] Fujimura J, Camilleri M, Low PA, Novak V, Novak P, Opfer-Gehrking TL. Effect of perturbations and a meal on superior mesenteric artery flow in patients with orthostatic hypotension. J Auton Nerv Syst. 1997 Dec 3;67(1-2):15-23. doi: 10.1016/s0165-1838(97)00087-8. PMID 9470140
- [Background] Chaudhuri KR, Thomaides T, Mathias CJ. Abnormality of superior mesenteric artery blood flow responses in human sympathetic failure. J Physiol. 1992 Nov;457:477-89. doi: 10.1113/jphysiol.1992.sp019388. PMID 1297840
- [Background] Tani H, Singer W, McPhee BR, Opfer-Gehrking TL, Haruma K, Kajiyama G, Low PA. Splanchnic-mesenteric capacitance bed in the postural tachycardia syndrome (POTS). Auton Neurosci. 2000 Dec 28;86(1-2):107-13. doi: 10.1016/S1566-0702(00)00205-8. PMID 11269915
- [Background] Revicki DA, Wood M, Wiklund I, Crawley J. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res. 1998 Jan;7(1):75-83. doi: 10.1023/a:1008841022998. PMID 9481153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started June 20, 2017. Participants were enrolled in Vanderbilt University medical center
Pre-assignment Details: We enrolled 26 subjects:
  * 25 subjects completed the study.
  * 1 subject was excluded from analysis because she was using GLP-1 agonist for weight control
Groups:
- POTS Subjects: Participants with postural orthostatic tachycardia syndrome diagnosis. Oral glucose tolerance test: 75 grams of glucose
- Healthy Controls: Healthy subjects Oral glucose tolerance test: 75 grams of glucose
Period: Overall Study
Arm/Group | POTS Subjects | Healthy Controls
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — 1 subject was excluded from analysis because she was using GLP-1 agonist for weight contro | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- POTS: Patients with postural orthostatic tachycardia syndrome diagnosis.
  Oral glucose tolerance test: 75 grams of glucose
- Total: Total of all reporting groups
Arm/Group | POTS | Healthy Controls | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.7) | 29.9 (7.8) | 33.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 168.4 (5.8) | 168.5 (5.3) | 168.4 (5.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.4 (4.1) | 22.5 (3.2) | 22.9 (3.6)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dl] | 90.2 (21.2) | 80.4 (12.6) | 85.3 (16.9)
Insulin [Mean (Standard Deviation); unit: mlU/ml] | 8.4 (2.8) | 7.5 (3.8) | 7.95 (3.3)
Hematocrit [Mean (Standard Deviation); unit: Percentage of RBC mass to original blood] | 38.3 (2.8) | 35.9 (2.2) | 37.1 (2.5)
Hemoglobin [Mean (Standard Deviation); unit: mg/dl] | 12.9 (1.2) | 12.1 (0.8) | 12.5 (1.0)
AST [Mean (Standard Deviation); unit: unit/L] | 22.6 (7.6) | 20.2 (5.3) | 21.4 (6.4)
ALT [Mean (Standard Deviation); unit: unit/L] | 16.1 (5.4) | 15.3 (9.7) | 15.7 (7.55)
Total Bilirubin [Mean (Standard Deviation); unit: mg/dl] | 0.5 (0.2) | 0.7 (0.5) | 0.6 (0.35)

OUTCOME MEASURES:

1. Primary Outcome: C-peptide Levels After Oral Glucose Tolerance Test
Description: The plasma levels of GIP (Glucose-dependent insulinotropic polypeptide) ,GLP-1, C-peptide, insulin) and their pattern of secretion after ingestion of 75 g glucose.
  C peptide measured in pg/ml
Time Frame: 0-120 minutes during intervention
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- C Peptide Level in POTS Patients: Participants with postural orthostatic tachycardia syndrome diagnosis. C peptide level after ingesting 75 grams of glucose at 120 mins
- C Peptide Level in Healthy Controls: Healthy subjects C peptide level after ingesting 75 grams of glucose at 120 mins
Arm/Group | C Peptide Level in POTS Patients | C Peptide Level in Healthy Controls
Number analyzed (Participants) | 12 | 13
pg/mL | 40.6 (9.5) | 23.2 (4.8)

2. Primary Outcome: Insulin Levels After Oral Glucose Tolerance Test
Description: The plasma levels of GIP (Glucose-dependent insulinotropic polypeptide) ,GLP-1, C-peptide, insulin) and their pattern of secretion after ingestion of 75 g glucose.
Time Frame: 0-120 minutes during intervention
Measure: Mean (Standard Deviation); unit: uU/mL
Groups:
- Insulin Levels in POTS Patients: Participants with postural orthostatic tachycardia syndrome diagnosis. Insulin levels after ingesting 75 grams of glucose at 120 mins
- Insulin Levels in Healthy Controls: Healthy subjects Insulin levels after ingesting 75 grams of glucose at 120 mins
Arm/Group | Insulin Levels in POTS Patients | Insulin Levels in Healthy Controls
Number analyzed (Participants) | 12 | 13
uU/mL | 85.2 (44.0) | 48.79 (13.69)

3. Primary Outcome: GIP and GLP-1 Levels After Oral Glucose Tolerance Test
Description: as for outcome 2
Time Frame: 0-120 minutes after the oral glucose ingestion
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- POTS Patients: Participants with postural orthostatic tachycardia syndrome diagnosis. GIP and GLP-1 levels after ingesting 75 grams of glucose at 120 mins
- Healthy Controls: Healthy subjects GIP and GLP-1 levels after ingesting 75 grams of glucose at 120 mins
Arm/Group | POTS Patients | Healthy Controls
Number analyzed (Participants) | 12 | 13
pmol/L
  GIP secretion at 120 mins | 75.72 (41.77) | 42.74 (9.6)
  GLP-1 secretion at 30 mins | 66.0 (23.0) | 53.9 (18.3)

4. Secondary Outcome: Changes in Systemic Hemodynamics After 75-gr Oral Glucose and During Orthostasis
Description: The percent change (before-after 75 gram of oral glucose) of standing heart rate and stroke volume (SV).
Time Frame: 0-120 mins
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | POTS | Healthy Controls
Number analyzed (Participants) | 12 | 13
Percent change
  % change in standing HR | 21.2 (11.9) | 6.0 (19.9)
  percent change in standing stroke volume | -10.3 (11.90) | 3.3 (13.7)

ADVERSE EVENTS:
Time Frame: At the time of study visit, up to 120 minutes
Arm/Group | POTS | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT03263819/Prot_SAP_000.pdf